CLINICAL TRIAL: NCT02424630
Title: The Effect of Sono-Guided Interscalene Brachial Plexus Block Combined With Arthroscopy-Guided Suprascapular Nerve Block in Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial
Brief Title: Interscalene Brachial Plexus Block Combined With Suprascapular Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Hallym University (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Assistant Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2013-52
Record Dates: First submitted 2015-04-17; First posted 2015-04-23 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Rotator Cuff Injury
Keywords: sono-guided interscalene brachial plexus block; arthroscopy-guided suprascapular nerve block; arthroscopic rotator cuff repair; postoperative pain
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ISB with SSNB (Experimental): During arthroscopic rotator cuff repair, ultrasound-guided ISB was performed preemptively with 7.5 mL ropivacaine immediately after general anesthesia was induced. And at the end of surgery, arthroscopy-guided SSNB was performed with 10 mL ropivacaine.
  Interventions: Device: Ultrasound-guided ISB; Device: Arthroscopy-guided SSNB; Drug: Placebo; Drug: Ropivacaine
- ISB alone (Placebo Comparator): During arthroscopic rotator cuff repair, ultrasound-guided ISB was performed preemptively with 7.5 mL ropivacaine immediately after general anesthesia was induced. And at the end of surgery, arthroscopy-guided SSNB was performed with 10 mL normal saline.
  Interventions: Device: Ultrasound-guided ISB; Drug: Placebo

INTERVENTIONS:
Device: Ultrasound-guided ISB — ISB was performed by one anesthesiologist under ultrasound-guidance. The superior, middle, and inferior trunks of the brachial plexus were identified approximately 2 cm above the clavicle. A 50 mm 22-gauge needle was introduced percutaneously using an out-of-plane technique. The needle was placed beside each trunk in succession, and 2.5 mL ropivacaine was injected into each site. The total volume of ropivacaine used for ISB was 7.5 mL.
Device: Arthroscopy-guided SSNB — At the end of the surgery, SSNB was performed under arthroscopic guidance by one shoulder arthroscopist. The suprascapular ligament was found using the lateral portal for visualization. The supraclavicular ligament was visualized at the end of the conoid ligament when the arthroscope was advanced following the coracoclavicular ligament. A 23-gauge spinal needle was introduced in a posteroanterior direction at a 20° angle percutaneously and 7 cm medial to the lateral margin of the acromion. Then, the needle was placed at the upper margin of the suprascapular ligament and advanced slightly under arthroscopy-guidance. After suctioning the saline from the portal, the injection material was administered according to the random assignment.
  Arms: ISB with SSNB
Drug: Placebo — All the regional blocks in this study were performed using ropivacaine, except for arthroscopy-guided SSNB using placebo (10 mL normal saline)
Drug: Ropivacaine — All the regional blocks in this study were performed using 10mL ropivacaine.
  Arms: ISB with SSNB

SUMMARY:
The investigators compared the results of sono-guided interscalene brachial plexus block (ISB) combined with arthroscopy-guided suprascapular nerve block (SSNB) with those of ISB alone within the first 48 h after arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
Forty-eight patients with rotator cuff tears who had undergone arthroscopic rotator cuff repair were enrolled. The 24 patients randomly allocated to group 1 received ISB and SSNB; the remaining 24 patients in group 2 underwent ISB alone. VAS pain score, patient's satisfaction (SAT) were checked postoperative 1, 3, 6, 12, 18, 24, 36, and 48 hours. VAS pain score was selected from 0 to 10 was no pain and 10 was severe pain that the patient had ever experienced. SAT was also selected from 0 to 10 was unsatisfactory and 10 was very satisfactory. Rebound of postoperative pain was confirmed if there had been an increase of VAS pain score after postoperative 1 hour.

ELIGIBILITY:
Inclusion Criteria:

1. definite rotator cuff tear on preoperative MRI, which needed repair;
2. acceptance of arthroscopic surgery including rotator cuff repair;
3. > 20 years old; and
4. acceptance of routine regional blocks and patient-controlled analgesia.

Exclusion Criteria:

1. did not want arthroscopic rotator cuff repair;
2. stopped PCA before 48 h postoperatively due to side effects;
3. history of shoulder operation or fracture;
4. concomitant neurological disorder around the shoulder;
5. conversion to open surgery from the arthroscopy; and
6. contraindication to the routine regional blocks in this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD, PhD, Principal Investigator — Chuncheon Sacred Heart Hospital

REFERENCES:
- [Derived] Lee JJ, Hwang JT, Kim DY, Lee SS, Hwang SM, Lee NR, Kwak BC. Effects of arthroscopy-guided suprascapular nerve block combined with ultrasound-guided interscalene brachial plexus block for arthroscopic rotator cuff repair: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Jul;25(7):2121-2128. doi: 10.1007/s00167-016-4198-7. Epub 2016 Jun 16. PMID 27311449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Rotator cuff tears were diagnosed by preoperative MRI, and the size of the rotator cuff was confirmed at the time of surgery. The indication for surgery was a symptomatic full thickness rotator cuff tear or a > 50% thickness partial thickness rotator cuff tear. From Aug 2013 to Jul 2014, the recruitment was done at Orthopeic department.
Pre-assignment Details: Assessed for eligibility (n= 54) Excluded (n= 2) previous fracture history of affected shoulder (n= 1) previous cerebral palsy history involving affected shoulder(n= 1) preassignment(n=52)
Groups:
- ISB With SSNB: During arthroscopic rotator cuff repair, ultrasound-guided ISB was performed preemptively with 7.5 mL ropivacaine immediately after general anesthesia was induced. And at the end of surgery, arthroscopy-guided SSNB was performed with 10 mL ropivacaine.
  Ultrasound-guided ISB: ISB was performed by one anesthesiologist under ultrasound-guidance. The superior, middle, and inferior trunks of the brachial plexus were identified approximately 2 cm above the clavicle. A 50 mm 22-gauge needle was introduced percutaneously using an out-of-plane technique. The needle was placed beside each trunk in succession, and 2.5 mL ropivacaine was injected into each site. The total volume of ropivacaine used for ISB was 7.5 mL.
  Arthroscopy-guided SSNB: At the end of the surgery, SSNB was performed under arthroscopic guidance by one shoulder arthroscopist.
Period: Overall Study
Arm/Group | ISB With SSNB | ISB Alone
Started | 25 | 27
Completed | 24 | 24
Not Completed | 1 | 3
Not completed — No rotator cuff tear | 1 | 2
Not completed — Open procedure | 0 | 1

BASELINE CHARACTERISTICS:
Population: A power analysis indicated that 44 patients (22 patients in each cohort) would provide a statistical power of 80% with a two-sided α-level of 0.05 to detect a significant difference in the VAS score 12 h postoperatively, assuming an effect size of 0.89 (mean difference, 1.6; standard deviation [SD], 1.8).
Groups:
- ISB Alone: During arthroscopic rotator cuff repair, ultrasound-guided ISB was performed preemptively with 7.5 mL ropivacaine immediately after general anesthesia was induced. And at the end of surgery, arthroscopy-guided SSNB was performed with 10 mL normal saline.
  Ultrasound-guided ISB: ISB was performed by one anesthesiologist under ultrasound-guidance. The superior, middle, and inferior trunks of the brachial plexus were identified approximately 2 cm above the clavicle. A 50 mm 22-gauge needle was introduced percutaneously using an out-of-plane technique. The needle was placed beside each trunk in succession, and 2.5 mL ropivacaine was injected into each site. The total volume of ropivacaine used for ISB was 7.5 mL.
  Placebo
- Total: Total of all reporting groups
Arm/Group | ISB With SSNB | ISB Alone | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.6) | 57.3 (12.0) | 57.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Score
Description: The VAS pain score was based on a scale from 0 to 10, where 0 indicated no pain and 10 indicated severe pain
Time Frame: 1, 3, 6, 12, 18, 24, 36, 48h
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ISB With SSNB | ISB Alone
Number analyzed (Participants) | 24 | 24
units on a scale
  1h | 2.0 (1.2) | 2.6 (1.4)
  3h | 1.7 (1.0) | 2.6 (1.4)
  6h | 1.6 (1.1) | 4.0 (2.2)
  12h | 3.5 (1.9) | 5.8 (1.5)
  18h | 3.6 (1.7) | 5.2 (1.6)
  24h | 3.2 (1.7) | 4.2 (1.5)
  36h | 2.1 (1.1) | 2.7 (1.0)
  48h | 1.3 (0.8) | 2.0 (0.7)

2. Secondary Outcome: Patient Satisfaction (SAT) Score
Description: The SAT score was also from 0 to 10, where 0 indicated unsatisfactory and 10 indicated very satisfactory.
Time Frame: 1, 3, 6, 12, 18, 24, 36, 48h
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ISB With SSNB | ISB Alone
Number analyzed (Participants) | 24 | 24
units on a scale
  1h | 7.9 (1.3) | 7.2 (1.4)
  3h | 7.8 (1.1) | 7.3 (1.4)
  6h | 7.8 (1.0) | 6.0 (1.9)
  12h | 6.2 (1.4) | 4.3 (1.4)
  18h | 6.4 (1.3) | 5.1 (1.5)
  24h | 6.9 (1.2) | 5.9 (1.7)
  36h | 7.9 (1.1) | 7.1 (1.2)
  48h | 8.5 (0.6) | 8.2 (0.9)

ADVERSE EVENTS:
Time Frame: During operation
Description: During operation, hypoxia was checked using arterial SaO2.
Arm/Group | ISB With SSNB | ISB Alone
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No